CLINICAL TRIAL: NCT01486992
Title: mFOLFIRI Combine With Nimotuzumab Second Line Chemotherapy for Squamous-cell Carcinoma of the Esophagus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, HEAD OF GI ONCOLOGY, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N+FOLFIRI-AEC-4
Record Dates: First submitted 2011-11-22; First posted 2011-12-07 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2011-11

CONDITIONS: Advanced Esophageal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nimotuzumab (Experimental): irinotecan 180mg/m2，iv ，d1，LV 200 mg/m2 ，2h，d1，5-FU 400 mg/m2， iv，d1 5-FU 2400mg/m2，CIV，46h，q2w Nimotuzumab 200mg，iv，qw
  Interventions: Drug: mFOLFIRI+Nimotuzumab

INTERVENTIONS:
Drug: mFOLFIRI+Nimotuzumab — irinotecan 180mg/m2，iv ，d1，LV 200 mg/m2 ，2h，d1，5-FU 400 mg/m2， iv，d1 5-FU 2400mg/m2，CIV，46h，q2w Nimotuzumab 200mg，iv，qw

SUMMARY:
There are few studies about 2nd line treatment in advanced esophageal carcinoma (AEC), some showed that irinotecan may be effective. The investigators previous study has shown the efficacy and safety of paclitaxel/cisplatin as 1st line treatment, so in this phase II study, the investigators would like to observe the efficacy and safety of Nimotuzumab plus Irinotecan/5FU/leucovorin as 2nd line treatment if AEC after failure to 1st treatment of PTX/DDP.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal squamous carcinoma,failed to 1st line treatment of paclitaxel/cisplatin
* Age 18 to 75 years old
* Measurable disease according to the RECIST criteria(diameter of the lesion should be more than 10mm by spiral CT or MRI, more than 20mm by common CT, the date of image should be less than 15 days before enrollment)
* Life expectancy of ≥3 month
* Karnofsky performance status ≥80
* WBC>3,500/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl，Bilirubin level < 1.0 times ULN，Serum creatinine <1.0 times ULN，ALT and AST<2.5 times ULN ，AKP < 2.5 times ULN ，(≤5 times ULN in patients with liver metastases)(within 7 days before enrollment)
* No sever complication, such as active gastrointestinal bleeding, perforation, jaundice, obstruction, non-cancerous fever>38℃；
* Normal ECG/cardiac function
* Good compliance
* Having signed informed consent

Exclusion Criteria:

* More than 1 Previous systemic therapy for metastatic esophageal squamous carcinoma
* Known hypersensitivity to study drugs
* Tumor with length≥10cm, liver metastasis covers more than 50% of liver,or lung metastasis covers more than 25% of lung
* No measurable lesions, eg. pleural fluid and ascites
* Only with Other previous malignancy within 5 year, except non-melanoma skin cancer
* Heart failure or other sever organ dysfunction, eg. coronary artery disease, myocardial infarction within the last 6 months only Brain or bone metastasis
* Chronic diarrhea
* Mentally abnormal or disable cognition,including CNS metastasis
* Pregnancy or lactation period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 years
adverse events | 2 weeks

SECONDARY OUTCOMES:
progression-free survival | 1year
response rate | 6 weeks
disease control rate | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhang Xiaodong, Beijing, Beijing Municipality, China